CLINICAL TRIAL: NCT04776954
Title: Comparison of Normothermia Maintenance Between Resistive Blanket and Forced Air Warming Systems in Renal Transplant Surgery
Brief Title: Warming Blanket Comparison Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left institution, no new PI available
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ANES-2021-29543
Record Dates: First submitted 2021-02-25; First posted 2021-03-02 (Actual); Results first posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Surgery; Temperature Change, Body
MeSH Terms: conditions — Body Temperature Changes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Forced Air Warming System (Active Comparator): Participants in this arm will receive warming using a forced air warming system.
  Interventions: Device: Forced Air Warming System
- Resistive Blanket Warming System (Active Comparator): Participants in this arm will receive warming using a resistive blanket warming system.
  Interventions: Device: Resistive Blanket Warming System

INTERVENTIONS:
Device: Forced Air Warming System — The forced air warming system has a heater unit that blows air through a conduit to an "air blanket" that inflates with forced air that circulates throughout the blanket, and exits through tiny perforations on the patient-side of that blanket. The heat primarily warms the subject through convective means. As the warmed air escapes through the perforations in the blanket, it creates an environment of continuously circulating warm air that is in contact with the skin.
  Arms: Forced Air Warming System
Device: Resistive Blanket Warming System — This blanket is equivalent to an operating-room-safe electric blanket. Through a power cord, a separate power source powers a semiconductor layer within the resistive blanket to generate heat. The heat primarily warms the subject by conductive warming through direct skin contact, and, secondarily, by warming the air around the participant in areas where there is no direct skin contact.
  Arms: Resistive Blanket Warming System

SUMMARY:
The purpose of the study is to compare the effectiveness of resistive blanket warming to forced air warming in maintaining body temperature in participants undergoing renal transplantation.

DETAILED DESCRIPTION:
The study will involve two arms: a resistive blanket warming system arm and a forced air warming system arm. Both devices will be set to warm the participant at a standard 41 degrees Celsius when the participant is to be rewarmed.

During the study, the forced air warming system (FAWS) will be placed on the (resistive blanket warming system (RBWS), with the participant laying on top of the forced air warming system. The arm components will be wrapped around the participant's arms to assist with patient positioning for surgery. Both the forced air and resistive blanket warming systems will be attached to their respective heating units before the participant is brought to the OR and transferred to the operating room table. After the needed standard monitors for surgery have been placed, general anesthesia will be induced and maintained with participant's hemodynamics and other vitals maintained per standard care (no additional measurements beyond standard of care which is recorded in EPIC). The certified registered nurse anesthetists (CRNA) will be involved in the placement of the blankets. Operating Room Nurse managers and CRNA's will be informed by research team regarding participant's involvement in the study.

Participant's core temperature will be measured with a nasopharyngeal temperature probe. Vital signs, including continuous blood pressure, heart rate, oxygen saturation, and end-tidal carbon dioxide, will be monitored and recorded in Epic as is routine with all anesthetics performed.

Standard anesthetic care of the participant will occur for the duration of the surgery. The participant will be randomized to either the FAWS or RBWS before arrival to the operating room. The participant's temperature will be monitored and recorded for the duration of surgery with the selected warming system. The primary outcome variable is the nasopharyngeal temperature as recorded at the end of the surgery.

Temperature measurement in the PACU will be standardized with skin temperature probes that will be placed on the forehead prior to leaving the operating room.

ELIGIBILITY:
Inclusion Criteria:

- Undergoing elective renal transplantation

Exclusion Criteria:

* Previous surgery involving organ transplantation or nephrectomy. These patients are at higher risk of blood loss, making temperature regulation subject to more variables outside our control.
* End stage renal disease with decreased or no urine output from normal. Bladder temperature will not be valid in these patients.
* Previous upper extremity amputations
* Ongoing sepsis or other infection
* Thyroid dysfunction
* Emergency surgery
* Refusal of consent to participate in study
* Pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2022-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cole Bennett, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Forced Air Warming System | Resistive Blanket Warming System
Started | 7 | 8
Completed | 7 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Forced Air Warming System | Resistive Blanket Warming System | Total
Number analyzed (Participants) | 7 | 8 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 6 | 11
  >=65 years | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 6 | 4 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 12
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 6 | 7 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: AUC of Temperature vs Time
Description: Outcome is reported as the Area Under Curve (AUC) of temperature vs time curve during hypothermia (core temperature less than 36 degrees Celcius) during the duration of surgery. Unit of measure is degrees Celsius per minute.
  Time during surgery spent under 36 degrees Celsius through comparison of nasopharyngeal temperature, which is measured by placing a nasopharyngeal temperature probe 10 to 20 cm into the nare, between forced air warming system (FAWS) and resistive blanket warming system (RBWS).
Time Frame: up to 5 hours
Measure: Mean (Standard Deviation); unit: celsius per minute
Arm/Group | Forced Air Warming System | Resistive Blanket Warming System
Number analyzed (Participants) | 7 | 8
celsius per minute | -131 (93) | -147 (69)

2. Secondary Outcome: Body Temperature Upon Arrival in PACU
Description: Outcome is reported as the body temperature recorded upon arrival in post-anesthesia care unit (PACU).
Time Frame: up to 2 hours
Measure: Mean (Standard Deviation); unit: celsius per minute
Arm/Group | Forced Air Warming System | Resistive Blanket Warming System
Number analyzed (Participants) | 7 | 8
celsius per minute | 36.8 (0.5) | 37 (0.3)

ADVERSE EVENTS:
Time Frame: No adverse event were reported. The study participants were only on the study for the time of warming blanket and was very minimal risk.
Description: No AE data collected during the study
Arm/Group | Forced Air Warming System | Resistive Blanket Warming System
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-06): https://cdn.clinicaltrials.gov/large-docs/54/NCT04776954/Prot_SAP_000.pdf
  • Informed Consent Form (2022-02-23): https://cdn.clinicaltrials.gov/large-docs/54/NCT04776954/ICF_001.pdf